CLINICAL TRIAL: NCT02066467
Title: Maximizing CRT Delivery by Using Multipolar Coronary Sinus Lead Family ACUITY® X4
Brief Title: Maximizing CRT Delivery by Using MultipolAr Coronary Sinus Lead FamiLy ACUITY® X4 - RALLY X4 Study
Acronym: RallyX4
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Other Study IDs: Rally X4-10-2013
Record Dates: First submitted 2014-02-07; First posted 2014-02-19 (Estimated); Results first posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-08

CONDITIONS: Heartfailure
Keywords: Phrenic Nerve Stimulation; Heartfailure treatment; CRT-D therapy; Quadripolar lead; Lead related complication free rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart failure patients: * Subjects with art failure who receive stable optimal pharmacologic therapy
  * Moderate to severe heart failure (NYHA Class III-IV) with ejection fraction (EF) ≤ 35% and QRS duration ≥ 120 ms
  * Left bundle branch block (LBBB) with QRS duration ≥ 130 ms, EF ≤ 30%, and mild (NYHA Class II) ischemic or non-ischemic heart failure or asymptomatic (NYHA Class I) ischemic heart failure.
  The study is collecting observational data on regular CRT-D device implants with special focus on the left ventricular ACUITY X4® Lead Family' .
  Interventions: Device: Left Ventricular lead implant: ACUITY X4® Lead Family

INTERVENTIONS:
Device: Left Ventricular lead implant: ACUITY X4® Lead Family — Implantation of (cardiac re-synchronization therapy with defibrillator) CRT-D devices for heartfailure treatment
  Other Names: Autogen™X4 CRT-D G179-200 G177-200; Dynagen™ X4 CRT-D G158-200 G156-200; Inogen™ X4 CRT-D G148-200 G146-200; Origen™ X4 CRT-D G058-200 G056-200

SUMMARY:
The objective of this study is to collect clinical data on safety and performance of ACUITY X4® leads when used in a standard clinical setting.

It is a prospective, non-randomized, observational multicenter study evaluating standard of care.

For Post Market Clinical Follow up (PMCF) purposes the 3 month implant success rate, adverse events and basic parameters of the lead will be assessed. The cohort of subjects included in this evaluation will be the first 200 subjects which are indicated for PMCF in Rally X4 to receive an ACUITY X4® lead implant.

Study endpoints:

Phrenic Nerve Stimulation (PNS) related CFR through 6 months post-implant (Defined as: rate of freedom from loss of function or operative system revision due to unacceptable PNS threshold) Lead-related Complication-Free Rate (CFR) from Implant through 3 months post-implant.

DETAILED DESCRIPTION:
Clinic visits will occur at:

* Enrollment and Consenting Clinic Visit (≤ 30 days prior to implant procedure)
* Implant Procedure (Day 0; all future follow ups based on this date)
* Pre-Discharge Clinic Visit (≤ 7 days post implant procedure) (Required)
* One to 6 Month Clinic Visit (20 to 180 days post implant procedure) (Required)
* Interim Visit(s) (Any time between the 1 to 6 Month Clinic Visit and Close-out Clinic Visit) (Following study center specific standard of care) (Device follow up optional) AE - reporting required
* Close-out Clinic Visit (30 months ± 90 days, OR 180 days ± 90 days after the study is closed to enrollment, whichever comes first) (Required)
* During the trial all AEs, deaths, and changes in the device system must be reported
* Devices of subjects who have received a Latitude device will be followed by the Boston Scientific (BSC) Latitude team. Device Data as defined in the Clinical Investigation Plan (CIP), device alerts, and diagnostic data from the standard Latitude database may be collected and entered into the study database at any time.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and capable of providing informed consent
2. Subject is planned to be implanted with an ACUITY X4® lead for left-ventricular pacing and sensing via the coronary venous system in conjunction with a compatible BSC pulse generator
3. Subject is willing and capable of participating in all visits associated with this study at an approved clinical study center and at the intervals defined by this CIP
4. Subject is age 18 or above, or of legal age to give informed consent specific to state and national law

Exclusion Criteria:

1. Subjects with a hypersensitivity to a maximum single dose of 0.51 mg dexamethasone acetate
2. Subject is enrolled in any other concurrent study without prior written approval from BSC, with the exception of local mandatory governmental registries and observational studies/registries that are not in conflict and do not affect the following:

   * Schedule of procedures for the RALLY X4 Study (i.e. should not cause additional or missed visits);
   * RALLY X4 Study outcome (i.e. involve medications that could affect the heart rate of the subject);
   * Conduct of the RALLY X4 Study per GCP/ ISO 14155:2011/ local regulations as applicable
3. Per the implanting physician's discretion, the subject is not a suitable candidate to receive the study device as determined during the implant procedure
4. Women of childbearing potential who are or might be pregnant at the time of study enrollment or ACUITY X4® lead implant.
5. Subject is unwilling or unable to participate in all scheduled study follow up visits at an approved study center
6. Subject does not anticipate being a resident of the area for the scheduled duration of the trial
7. Subject's physician does not allow participation

   -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The BSC Cardiac Resynchronization Therapy Defibrillators (CRT-Ds) are indicated for subjects with art failure who receive stable optimal pharmacologic therapy (OPT) for heart failure and who meet any one of the following classifications:
  * Moderate to severe heart failure (New York Heart Association (NYHA) Class III-IV) with ejection fraction (EF) ≤ 35% and QRS duration ≥ 120 ms
  * Left bundle branch block (LBBB) with QRS duration ≥ 130 ms, EF ≤ 30%, and mild (NYHA Class II) ischemic or non-ischemic heart failure or asymptomatic (NYHA Class I) ischemic heart failure BSCCRT-Ds are also intended to provide ventricular antitachycardia pacing and ventricular defibrillation for automated treatment of life-threatening ventricular arrhythmias.
Sampling Method: Non-Probability Sample
Enrollment: 863 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haran Burri, Prof., Principal Investigator — Hôpital Cantonal de Genève; Torsten Kayser, Study Chair — Boston Scientific Corporation
Locations (83):
- Landesklinikum St.Pölten, Sankt Pölten, Austria
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Guidant Europe SA / NV a Boston Scientific Company, Diegem
  - Universitair Ziekenhuis Gent, Ghent
- Colombia (3):
  - Fundation Cardioinfantil, Bogotá
  - Fundación Valle del Lili, Cali
  - Clinica Medellin, Medellín
- Denmark (2):
  - Gentofte Hospital, Copenhagen
  - Aarhus University Hospital, Skejby
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Oulu University Hospital, Oulu
- France (11):
  - CHU Amiens, Amiens
  - Centre Hospitalier d'Annecy, Annecy
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Hôpital de la Timone, Marseille
  - Nouvelles Cliniques Nantaises, Nantes
  - Centre Hospitalier de Pau, Pau
  - CHU de Rennes, Rennes
  - CH de Rouen, Rouen
  - Clinique Pasteur, Toulouse
- Germany (9):
  - Herzzentrum Nordrhein-Westfalen, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin, Berlin
  - Unfallkrankenhaus Berlin, Berlin
  - Waldklinikum Gera, Gera
  - Herz-und Gefäßzentrum Göttingen, Göttingen
  - Klinikum Kassel, Kassel
  - Krankenhaus Landshut-Achdorf, Landshut
  - University Magdeburg, Magdeburg
  - Klinikum Oldenburg, Oldenburg
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Waterfort Hospital, Waterford, Ireland
- Israel (5):
  - Barzilai Medical Center, Ashkelon
  - Beilinson Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Medical Center, Tel Aviv
- Italy (8):
  - Policlinico Sant'Orsola-Malpighi, Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Policlinico Vittorio Emanuele, Catania
  - Ospedale Pugliese Ciaccio, Catanzaro
  - Azienda Ospedaliera Spedale Sant'Anna di Como, Como
  - Clinica Montevergine, Mercogliano
  - Ospedale Santa Maria Misericordia, Rovigo
  - Ospedale Borgo Trento, Verona
- Japan (11):
  - Kansai Rosai Hospital, Amagasaki-Shi
  - Tokai University Hospital, Isehara-Shi
  - Shonan Kamakura General Hospital, Kamakura-Shi
  - Kokura Memorial Hospital, Kitakyushu-Shi
  - Kyorin University Hospital, Mitaka-Shi
  - Osaka General Medical Center, Osaka
  - Osaka Police Hospital, Osaka
  - Sakurabashi Watanabe Hospital, Osaka
  - Osaka Rosai Hospital, Sakaishi
  - Osaka University Hospital, Suita-Shi
  - Yokohama City University Hospital, Yokohama
- Netherlands (4):
  - Medisch Centrum Alkmaar, Alkmaar
  - Hospital Rijnstate, Arnhem
  - Medisch Spectrum Twente, Enschede
  - Isala, Zwolle
- Portugal (5):
  - Centro Hospitalar de Vila Nova de Gaia, Gaia
  - Centro Hospitalar do Alto Ave, Guimarães
  - Hospital Santa Cruz, Lisbon
  - Hospital Santa Maria, Lisbon
  - Centro Hospitalar do Porto, Porto
- Singapore (2):
  - Changi General Hospital, Singapore
  - National Heart Centre, Singapore
- Spain (7):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Sant Pau, Barcelona
  - Doce De Octubre University Hospital, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Vírgen de la Salud, Toledo
  - Hospital Clinico Valladolid, Valladolid
- Switzerland (3):
  - Hôpital Cantonal de Genève, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Institution Kantonsspital St. Gallen, Sankt Gallen
- United Kingdom (4):
  - Queen Elisabeth Hospital, Birmingham
  - Golden Jubilee National Hospital, Glasgow
  - Imperial College Healthcare, London
  - St Bartholomew's Hospital, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on 10 February 2014. The clinical phase of the study was completed on 30 September 2016 which was the date of the last subject's close-out visit. A total of 863 subjects across 82 centers were enrolled in the study in Europe, Asia and South America.
Groups:
- Heart Failure Patients: * Subjects with heart failure who receive stable optimal pharmacologic therapy
  * Moderate to severe heart failure (NYHA Class III-IV) with ejection fraction (EF) ≤ 35% and QRS duration ≥ 120 ms
  * Left bundle branch block (LBBB) with QRS duration ≥ 130 ms, EF ≤ 30%, and mild (NYHA Class II) ischemic or non-ischemic heart failure or asymptomatic (NYHA Class I) ischemic heart failure.
  The study is collecting observational data on regular CRT-D device implants with special focus on the left ventricular ACUITY X4® Lead Family' .
  Left Ventricular lead implant: ACUITY X4® Lead Family: Implantation of (cardiac re-synchronization therapy with defibrillator) CRT-D devices for heartfailure treatment
Period: Overall Study
Arm/Group | Heart Failure Patients
Started | 863
Completed | 648
Not Completed | 215
Not completed — Did not undergo implant procedure | 24
Not completed — Attempted to implant withoput success | 43
Not completed — Consent ineligible | 1
Not completed — Death | 54
Not completed — Lost to Follow-up | 51
Not completed — Adverse Event | 20
Not completed — Withdrawal by Subject | 16
Not completed — Physician Decision | 2
Not completed — Not defined | 4

BASELINE CHARACTERISTICS:
Arm/Group | Heart Failure Patients
Number analyzed (Participants) | 863
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189
  Male | 674
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Colombia | 13
  Singapore | 18
  Hong Kong | 9
  Japan | 60
  United Kingdom | 38
  Switzerland | 31
  Portugal | 33
  Spain | 67
  Austria | 15
  Netherlands | 57
  Belgium | 5
  Ireland | 12
  Finland | 23
  Denmark | 30
  Italy | 124
  Israel | 47
  France | 119
  Germany | 162

OUTCOME MEASURES:

1. Primary Outcome: Phrenic Nerve Complication Free Rate
Description: The Phrenic Nerve Stimulation (PNS) related Complication Free rate (CFR) through 6 months post-implant is defined as the rate of freedom from loss of function or operative system revision due to unacceptable PNS threshold
Time Frame: 6 months post-implant
Population: 795 patients successfully implanted with ACUITY X4 lead
Measure: Number (90% Confidence Interval); unit: % of participants
Arm/Group | Heart Failure Patients
Number analyzed (Participants) | 795
% of participants | 99.5 [98.8 to 99.8]
Statistical Analysis 1: Comparison: Heart Failure Patients; Test type: Other; p < 0.0001, exact binominal methodology

2. Secondary Outcome: 3 Month Lead-related Complication-Free Rate (CFR)
Description: Lead-related Complication-Free Rate (CFR) from implant through 3 months post-implant. Lead-related complications associated with the ACUITY X4® lead were counted towards this endpoint.
Time Frame: 3 months post-implant
Population: 795 patients successfully implanted with ACUITY X4 lead
Measure: Number (90% Confidence Interval); unit: % of participants
Arm/Group | Heart Failure Patients
Number analyzed (Participants) | 795
% of participants | 98.8 [98 to 99.3]

3. Other Pre Specified Outcome: 3 Month Implant Success Rate for Indicated Subjects
Description: Post Market Clinical Follow-up (PMCF) of the ACUITY X4® lead was evaluated in this study. The outcome of interest is the 3 month implant success rate. The cohort of subjects included in this evaluation is the first 200 subjects to receive an ACUITY X4® lead implant and meet the PMCF eligibility criteria outlined below. The outcomes of interest for the PMCF supplemental analysis is the percent of subjects successfully implanted with an ACUITY X4® lead.
  Implant success is defined as the ability of the ACUITY X4® lead to be implanted and deliver CRT therapy. Subjects who have multiple lead implant attempts during the procedure, but are eventually successfully implanted with the ACUITY X4® lead and receive CRT therapy are classified as a successful implant.
Time Frame: 3 months post-implant
Population: At data cutoff date on 16 November 2015, 201 enrolled subjects met all of the PMCF eligibility criteria and were included in the analysis.
Measure: Number (90% Confidence Interval); unit: % of participants
Arm/Group | Heart Failure Patients
Number analyzed (Participants) | 201
% of participants | 99.5 [97.7 to 100]
Statistical Analysis 1: Comparison: Heart Failure Patients; Test type: Other; p < 0.0001, exact binominal methodology

ADVERSE EVENTS:
Time Frame: Adverse events are collected from 1st enrollment through study completion (last subject's close-out visit)
Description: All adverse events are collected as per ISO 14155:2011 and medical device guidance (MEDDEV) 2.7/3 12/2010 The number of participants at risk is defined as the subjects actively enrolled (838). Adverse events were not collected for subjects who did not undergo an implant procedure (24) and consent ineligible subjects (1).
Arm/Group | Heart Failure Patients
All-Cause Mortality (participants affected / at risk) | 54/838
Serious Adverse Events (participants affected / at risk) | 338/838
Other Adverse Events (participants affected / at risk) | 452/838
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heart Failure Patients (N=838)
Abnormal laboratory values (General disorders) | 2 (2)
Adverse reaction - Allergic reaction (General disorders) | 1 (1)
Adverse reaction - Hypotension (General disorders) | 1 (1)
Aortic regurgitation (Cardiac disorders) | 1 (1)
Aortic stenosis (Cardiac disorders) | 1 (1)
Arterial/venous thrombolytic event (Vascular disorders) | 1 (1)
Atrial fibrillation (AF) (Cardiac disorders) | 41 (46)
Atrial flutter (Cardiac disorders) | 10 (11)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (9)
Cardiac arrest (Cardiac disorders) | 3 (3)
Cardiogenic shock (Cardiac disorders) | 4 (5)
Cerebrovascular accident (CVA) (Cardiac disorders) | 5 (5)
Chest pain - Ischemic (Cardiac disorders) | 5 (6)
Chest pain - Other (Cardiac disorders) | 6 (7)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Coronary Artery Disease (Cardiac disorders) | 6 (6)
Coronary venous dissection (Surgical and medical procedures) | 1 (1)
Death (General disorders) | 13 (13)
Device Deficiency (Product Issues) | 1 (1)
Dislodgment - Elevated threshold - LV (Product Issues) | 1 (1)
Dislodgment - Extracardiac stimulation- LV (Product Issues) | 2 (2)
Dislodgment - Multiple signs - LV (Product Issues) | 1 (1)
Dislodgment - No reported signs - RA (Product Issues) | 4 (4)
Dislodgment - No reported signs - RV (Product Issues) | 3 (3)
Dislodgment - No reported signs -LV (Product Issues) | 2 (2)
Dislodgment - Unable to capture - LV (Product Issues) | 2 (2)
Dislodgment - Unable to capture - RA (Product Issues) | 1 (1)
Dislodgment - Unable to capture - RV (Product Issues) | 2 (2)
Distal thromboemboli (Cardiac disorders) | 1 (1)
Dizziness (Cardiac disorders) | 1 (1)
Dyspnea (Cardiac disorders) | 3 (3)
Dyspnea - Heart failure (Cardiac disorders) | 9 (11)
Elevated threshold - LV (Product Issues) | 4 (4)
Elevated threshold - RV (Product Issues) | 2 (2)
Endocrine (Endocrine disorders) | 3 (3)
Erosion (Product Issues) | 1 (1)
Extracardiac stimulation - LV (Product Issues) | 4 (4)
Extracardiac stimulation - RV (Product Issues) | 1 (1)
Fatigue (Cardiac disorders) | 1 (1)
Fever (Infections and infestations) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 20 (24)
Genitourinary (Reproductive system and breast disorders) | 4 (5)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 10 (11)
Heart failure symptoms - Unspecified (Cardiac disorders) | 49 (56)
Hematological (Blood and lymphatic system disorders) | 4 (5)
Hematoma - Pocket (<= 30 days post-implant) (Surgical and medical procedures) | 8 (8)
Hypertension (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Immune (Immune system disorders) | 2 (2)
Impedance > 2000 ohms - LV (Product Issues) | 1 (1)
Inappropriate tachy therapy - Noise (Product Issues) | 1 (1)
Inappropriate tachy therapy - Other (Product Issues) | 1 (1)
Inappropriate tachy therapy - SVT (Product Issues) | 6 (6)
Inappropriate tachy therapy- NSR (Product Issues) | 1 (1)
Infection (> 30 days post-implant) (Product Issues) | 10 (10)
Integumentary (Skin and subcutaneous tissue disorders) | 6 (8)
Intermittent Claudication (General disorders) | 1 (1)
Mitral regurgitation (Cardiac disorders) | 2 (2)
Mitral stenosis (Cardiac disorders) | 1 (1)
Multiple heart failure symptoms (Cardiac disorders) | 9 (10)
Multi-system failure (General disorders) | 3 (3)
Multi-system failure - Heart failure (Cardiac disorders) | 5 (5)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 9 (10)
Myocardial infarction (Cardiac disorders) | 3 (3)
Myocardial perforation post-implant - RA (Product Issues) | 1 (1)
Myocardial perforation post-implant - RV (Product Issues) | 4 (4)
Myocardial perforation with tamponade (Surgical and medical procedures) | 1 (1)
Myocardial perforation without tamponade (Surgical and medical procedures) | 1 (1)
Neurological (Nervous system disorders) | 3 (3)
Nonsustained ventricular tachycardia (NSVT) (Cardiac disorders) | 2 (2)
Other - Lead (Product Issues) | 7 (7)
Other - Lead - Procedure (Surgical and medical procedures) | 9 (9)
Other - PG system (Product Issues) | 1 (1)
Other - PG system - Procedure (Surgical and medical procedures) | 2 (2)
Other- Heart failure patient condition - Cardiovascular (Cardiac disorders) | 10 (12)
Other- Patient condition - Non- cardiovascular (General disorders) | 4 (4)
Other SVT (eg AVRT, AVNRT, EAT) (Cardiac disorders) | 5 (5)
Oversensing - RV (Product Issues) | 1 (1)
Pacemaker-mediated tachycardia (PMT) (Product Issues) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 3 (3)
Peripheral edema - Heart failure (Cardiac disorders) | 1 (1)
Peripheral vascular disease (Cardiac disorders) | 6 (6)
Physical trauma (General disorders) | 5 (5)
Pleural effusion - Procedure (Surgical and medical procedures) | 1 (1)
Pneumothorax - Procedure (Surgical and medical procedures) | 6 (6)
Post-surgical infection (<= 30 days post-implant) (Surgical and medical procedures) | 7 (8)
Post-surgical pocket hemorrhage (Surgical and medical procedures) | 2 (2)
Post-surgical wound discomfort (Surgical and medical procedures) | 1 (1)
Premature ventricular contractions (PVC) (Cardiac disorders) | 2 (2)
Psychological (Psychiatric disorders) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 23 (28)
Pulmonary edema - Heart failure (Cardiac disorders) | 2 (3)
Pulmonary embolism (PE) (Cardiac disorders) | 2 (2)
Renal (Renal and urinary disorders) | 12 (12)
Renal insufficiency - Heart failure (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Syncope (Cardiac disorders) | 1 (1)
Systemic infection (Infections and infestations) | 3 (3)
Thromboembolic events (Cardiac disorders) | 1 (1)
Transient ischemic attack (TIA) (Cardiac disorders) | 1 (1)
Unable to capture - RA (Product Issues) | 1 (1)
Venous occlusion (Surgical and medical procedures) | 1 (1)
Ventricular fibrillation (VF) (Cardiac disorders) | 10 (15)
Ventricular tachycardia (VT) (Cardiac disorders) | 17 (27)
Weight gain - Heart failure (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heart Failure Patients (N=838)
Abnormal laboratory values (General disorders) | 3 (3)
Adverse reaction - General (General disorders) | 2 (2)
Adverse reaction - Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic regurgitation (Cardiac disorders) | 1 (2)
Atrial fibrillation (AF) (Cardiac disorders) | 30 (33)
Atrial flutter (Cardiac disorders) | 2 (2)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chest pain - Heart failure (Cardiac disorders) | 2 (2)
Chest pain - Ischemic (Cardiac disorders) | 2 (2)
Chest pain - Other (Cardiac disorders) | 5 (5)
Coronary venous dissection (Surgical and medical procedures) | 8 (8)
Device Deficiency (Product Issues) | 33 (41)
Dislodgment - Elevated threshold - LV (Product Issues) | 2 (2)
Dislodgment - Elevated threshold -RV (Product Issues) | 1 (1)
Dislodgment - Multiple signs - LV (Product Issues) | 1 (1)
Dislodgment - No reported signs - RV (Product Issues) | 1 (1)
Dislodgment - No reported signs -LV (Product Issues) | 1 (1)
Dislodgment - Unable to capture - LV (Product Issues) | 1 (1)
Dislodgment - Unable to capture - RA (Product Issues) | 1 (1)
Dislodgment - Undersensing - RV (Product Issues) | 1 (1)
Dizziness (Cardiac disorders) | 5 (5)
Dyspnea (Cardiac disorders) | 1 (1)
Dyspnea - Heart failure (Cardiac disorders) | 11 (13)
Elevated threshold - LV (Product Issues) | 13 (14)
Elevated threshold - RA (Product Issues) | 4 (5)
Elevated threshold - RV (Product Issues) | 4 (4)
Endocrine (Endocrine disorders) | 5 (5)
Extracardiac stimulation - LV (Product Issues) | 47 (55)
Extracardiac stimulation - RV (Product Issues) | 2 (3)
Fever (Infections and infestations) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 8 (8)
Genitourinary (Reproductive system and breast disorders) | 5 (5)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 10 (11)
Heart failure symptoms - Unspecified (Cardiac disorders) | 2 (4)
Hematological (Blood and lymphatic system disorders) | 2 (2)
Hematoma - Pocket (<= 30 days post-implant) (Surgical and medical procedures) | 13 (13)
Hematoma - Pocket (> 30 days post-implant) (Surgical and medical procedures) | 1 (1)
Hematoma - Unrelated to procedure or device (Cardiac disorders) | 1 (1)
Hypertension - Heart failure (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 3 (3)
Hypotension - Heart failure (Cardiac disorders) | 1 (1)
Impedance > 2000 ohms - LV (Product Issues) | 1 (1)
Impedance > 2000 ohms - RA (Product Issues) | 1 (1)
Impedance > 2000 ohms - RV (Product Issues) | 1 (1)
Inappropriate AV delay (Product Issues) | 1 (1)
Inappropriate tachy therapy - Other (Product Issues) | 1 (1)
Inappropriate tachy therapy - SVT (Product Issues) | 5 (5)
Infection (> 30 days post-implant) (Product Issues) | 2 (2)
Integumentary (Skin and subcutaneous tissue disorders) | 4 (4)
Multiple heart failure symptoms (Cardiac disorders) | 2 (2)
Multiple symptoms (Cardiac disorders) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 10 (12)
Neurological (Nervous system disorders) | 2 (2)
Nonsustained ventricular tachycardia (NSVT) (Cardiac disorders) | 3 (3)
Other - Lead (Product Issues) | 4 (4)
Other - Lead - Procedure (Surgical and medical procedures) | 87 (92)
Other - PG system (Product Issues) | 1 (1)
Other - PG system - Procedure (Surgical and medical procedures) | 10 (10)
Other- Heart failure patient condition - Cardiovascular (Cardiac disorders) | 1 (1)
Other- Patient condition - Non- cardiovascular (General disorders) | 1 (1)
Other SVT (eg AVRT, AVNRT, EAT) (Cardiac disorders) | 3 (3)
Oversensing - RV (Product Issues) | 1 (1)
Pacemaker-mediated tachycardia (PMT) (Product Issues) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pericarditis - Unrelated to procedure or device (Cardiac disorders) | 1 (1)
Peripheral edema - Heart failure (Cardiac disorders) | 3 (3)
Physical trauma (General disorders) | 1 (1)
Pleural effusion - Procedure (Surgical and medical procedures) | 1 (1)
Pneumothorax - Procedure (Surgical and medical procedures) | 2 (2)
Post-surgical wound discomfort (Surgical and medical procedures) | 6 (6)
Premature ventricular contractions (PVC) (Cardiac disorders) | 14 (16)
Psychological (Psychiatric disorders) | 2 (4)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Rate response inappropriate (Product Issues) | 1 (1)
Renal (Renal and urinary disorders) | 2 (2)
RVAT Communication (Product Issues) | 6 (6)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Syncope (Cardiac disorders) | 1 (1)
Thromboembolic events (Cardiac disorders) | 1 (1)
Transient ischemic attack (TIA) (Cardiac disorders) | 1 (1)
Unable to capture - LV (Product Issues) | 1 (1)
Vasovagal reaction (Cardiac disorders) | 1 (1)
Venous occlusion (Surgical and medical procedures) | 1 (1)
Ventricular fibrillation (VF) (Cardiac disorders) | 4 (4)
Ventricular tachycardia (VT) (Cardiac disorders) | 9 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. The sponsor can request changes to the communication.